CLINICAL TRIAL: NCT05535426
Title: A Prospective Human Clinical Study to Assess Primary Stability and Change in Stability by Resonance Frequency Analysis of Immediately Inserted and Restored Dental Implants Using pH-Modified Tetranite® Implant Stabilization Material
Brief Title: Feasibility Study to Assess Outcomes of Immediately Inserted and Restored Dental Implants Using pH-modified Tetranite
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: RevBio (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DVAL 22004
Record Dates: First submitted 2022-09-07; First posted 2022-09-10 (Actual); Last update posted 2022-10-26 (Actual); Status verified 2022-10

CONDITIONS: Adhesive Dental
Keywords: dental implant; stabilization; resonance frequency analysis (RFA); bone adhesive; implant success; bone height; primary stability

STUDY DESIGN:
Intervention Model Description: Single arm, objective performance criteria study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Tetranite Stabilized Dental Implants with Provisional Crown (Experimental): Extraction of maxillary anterior teeth followed by immediate insertion and stabilization of dental implants with Tetranite in otherwise non-stable sites. A provisional crown will also be inserted during this surgery.
  Interventions: Device: Tetranite Implant Stabilization Material

INTERVENTIONS:
Device: Tetranite Implant Stabilization Material — Dental adhesive for increased implant stabilization

SUMMARY:
The aim of this Pilot Study is to demonstrate the safety and efficacy of the use of Tetranite Implant Stabilization Material (TN-ISM) in delivering enhanced stability to immediately restored dental implants inserted into fresh extraction sockets, with both clinical and patient-related successful outcomes.

DETAILED DESCRIPTION:
The purpose of the present study is to evaluate the safety and efficacy of a single stage approach using Tetranite Implant Stabilization Material (TN-ISM). The purpose of the efficacy component of this study is a composite comprising: (1) First - To demonstrate and evaluate the ability of TN-ISM to achieve immediate implant stabilization in sites otherwise unable to provide primary stability without requiring the delay in treatment imposed by the current multi-staged standard-of-care method; (2) Second - To demonstrate and evaluate the ability of TN-ISM to achieve increasing short-term stabilization of implants as the device undergoes initial resorption and replacement with new bone; (3) Third - To demonstrate the ability of TN-ISM to aid in the maintenance of alveolar ridge contours without buccal plate collapse and loss of crestal bone height; and Fourth (4) - To demonstrate and evaluate the ability of a TN-ISM stabilized implant to achieve implant success (after criteria of Buser, et. al 1) after 12 months in situ while the device undergoes significant resorption, facilitates osteoconduction, and replacement with new bone. In addition to the Primary Endpoints of establishing the Safety and Efficacy of Implant Stabilization and Implant Success throughout the initial 12 months of post-implant and device placement, the study also assesses several secondary endpoints over the course of the study and one-year follow-up, as outlined in the sections below. These include assessment of incidence, duration, and severity of adverse effects and events; assessment of increasing implant stiffness; assessment of bone levels, bone volumetric changes; patient satisfaction surveys, and assessment of periodontal and peri-implant health integral to implant success.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must have voluntarily signed the informed consent form before any study related procedures;
* Subjects must be males or females who are a minimum of 20 years of age;
* Subjects who require a single anterior maxillary tooth extraction and desire a replacement with a dental implant and immediate temporary crown. Candidate subjects may require more than one extraction, and all sitesbut only one site will be considered for inclusion in the study;
* Subjects must have opposing dentition (natural teeth, fixed or removable restorations);
* Subjects must be committed to the study and the required follow-up visits;
* Subjects must be American Society of Anesthesiology Grade (ASA) I or ASA II;
* Subjects who present with a sound bony housing with a visible buccal plate evident at the crest and fenestrations limited to <5.0mm diameter on a cone beam CT;
* Subjects who present with a sound bony housing with a visible buccal plate evident at the crest and dehiscences limited to <3.0mm in any direction on a cone beam CT;
* There must be sufficient bone height crestal to critical anatomical structures, i.e., the piriform foramen, and maxillary sinus, to safely place a dental implant within the bone contours. Extraction sockets should be able to accommodate an implant ≥9.0mm in length;
* Anatomical conditions must be present to allow an implant crown restoration to be placed at the candidate site, e.g., sufficient interocclusal space, incisal Class1 or Class 2 Div 1 relation, appropriate angulation of the ridge, etc.

Exclusion Criteria:

* There is at least 2mm of apical bone below the apex of the extraction socket for positive seating of the implant;
* Any implant site in which placement of the selected implant leaves an (Horizontal Dimension of Defect) HDD > 2mm in the buccal direction between the implant surface and the labial plate at the most coronal aspect of the extraction socket.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2022-09-22 (Actual); Primary Completion 2024-03-01 (Estimated); Study Completion 2024-03-01 (Estimated)

PRIMARY OUTCOMES:
Implant Stabilization by Resonance Frequency Analysis | 12 months
  The primary endpoint is sufficient bone-to-implant interfacial stiffness post-placement of the implant stabilized by TN-ISM, whereby, sufficient bone-to-implant interfacial stiffness is measured by Resonance Frequency Analysis (RFA) expressed as mean Implant Stability Quotient (ISQ) at 12 months post TN-ISM device and implant placement. For the study to be considered successful, the lower bound of the one-sided 97.5% confidence interval for the mean ISQ should exceed the clinical threshold of 60.

SECONDARY OUTCOMES:
Implant Stabilization by Resonance Frequency Analysis | 15 minutes, 3 months, and 7 months
  Sufficient bone-to-implant interfacial stiffness measured by Resonance Frequency Analysis (RFA) expressed as Implant Stability Quotient (ISQ) at 15 minutes, 3 months, and 7 months post TN-ISM device and implant placement. For each timepoint to be considered successful, the lower bound of the one-sided 97.5% confidence interval for the mean ISQ should exceed the clinical threshold of 60;
Device Related Adverse Events | 12 months
  Low incidence, severity and duration of device-related adverse events throughout the 12 months post TN-ISM device and implant placement follow-up period
Implant Stabilization by Manual Palpation | 15 minutes, 1 month, 3 months, and 7 months
  Immediate implant stabilization demonstrated by lack of clinical mobility of the implant subjected to manual palpation in any direction at 15 minutes after application of the TN-ISM and at 1 month, 3 months and 7 months post TN-ISM device and implant placement;
Implant Success (Composite Measure) | 12 months
  Composite measure of implant success (after criteria of Buser1) at 12 months post TN-ISM device and implant placement consisting of:
  * Presence of the implant at its site of implantation; and,
  * Absence of a recurrent peri-implant infection with suppuration; and,
  * No perceptible mobility upon palpation;
  * Absence of encapsulation, defined as continuous radiolucency around the implant in a periapical radiograph
Volume Loss | 12 months
  Crestal bone level maintenance assessed by analysis of two-dimensional periapical radiographic records showing no more than a 1.0mm loss of height throughout the 12 months post TN-ISM device and implant placement follow-up period
Per-implant tissue health | 12 months
  Peri-implant tissue health demonstrated by direct measurement around the implant at 12 months post TN-ISM device and implant placement follow-up period as compared to existing conditions in the oral cavity near adjacent teeth to the implant site and to baseline around the implant at 3 months post placement
Patient Satisfaction | 12 months
  Subject satisfaction using the patient-reported outcome measures

CONTACTS AND LOCATIONS:
Locations (1):
- Norton Implants, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cochran DL, Jones A, Sugita R, Brown MC, Guda T, Prasad H, Ong JL, Pollack A, Kay GW. Immediate Dental Implant Stabilization in a Canine Model Using a Novel Mineral-Organic Adhesive: 4-Month Results. Int J Oral Maxillofac Implants. 2020 Jan/Feb;35(1):39-51. doi: 10.11607/jomi.7891. PMID 31923288